CLINICAL TRIAL: NCT03392961
Title: To Assess the Pharmacokinetics and Pharmacodynamics of IN-105 in Relation to the Pre-meal Dosing Time, Between-meal Interval and Type of Meal - A Phase 1, Three Cohort, Randomized, Placebo Controlled, Crossover Trial in Type 2 Diabetes Patients
Brief Title: Effect of Dosing Time and Meal on IN-105 (Insulin Tregopil) PK and PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN-105-DM-01-G-14
Record Dates: First submitted 2017-12-19; First posted 2018-01-08 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Oral insulin; Dosing time; Insulin concentration; Prandial insulin; Post Prandial Glucose (PPG)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 3 Cohorts Cohort 1: 5 periods, 4 treatments and 5 sequences with a partial replicate crossover design Cohort 2: 6 periods, 6 treatments and 6 sequences in a cross-over design Cohort 3: 6 periods, 6 treatments and 6 sequences in a cross over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IN-105 (Insulin Tregopil) (Experimental): Cohort1: Treatments A, B, and C: IN-105 administered at 30, 20 or 10 minutes before the ADA meal, respectively; Treatment D: Placebo administered at 20 minutes before the ADA meal.
  Cohort 2: Treatments A, B, and C: IN-105 administered at 4, 5, and 6 hours after the previous ADA meal, respectively; Treatments D, E, and F: Placebo administered at 4, 5, and 6 hours after the previous ADA meal, respectively.
  Cohort 3: For the first meal, IN-105 30 mg administered at the optimal pre meal time determined from Cohort 1 with ADA meal (Treatments A and D) or high fat meal (Treatments B and E) or high fiber meal (Treatments C or F).
  Interventions: Drug: IN-105 (Insulin Tregopil)
- Placebo tablet (Placebo Comparator): Cohort1: Treatments A, B, and C: IN-105 administered at 30, 20 or 10 minutes before the ADA meal, respectively; Treatment D: Placebo administered at 20 minutes before the ADA meal.
  Cohort 2: Treatments A, B, and C: IN-105 administered at 4, 5, and 6 hours after the previous ADA meal, respectively; Treatments D, E, and F: Placebo administered at 4, 5, and 6 hours after the previous ADA meal, respectively.
  Cohort 3: For the first meal, IN-105 30 mg administered at the optimal pre meal time determined from Cohort 1 with ADA meal (Treatments A and D) or high fat meal (Treatments B and E) or high fiber meal (Treatments C or F).
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: IN-105 (Insulin Tregopil) — 15 mg strength tablets for oral use used at a dose of 30 mg
  Arms: IN-105 (Insulin Tregopil)
Other: Placebo comparator — Placebo tablet for oral use
  Arms: Placebo tablet

SUMMARY:
A study to evaluate the PK and PD of oral IN-105 (Insulin Tregopil) w.r.t. time of dosing prior to meal, duration between meals and type of meal .

DETAILED DESCRIPTION:
A Phase 1, Randomized, Placebo Controlled, Crossover Trial in Type 2 Diabetes Patients to evaluate the effect of pre-meal dosing time, inter-meal interval and meal composition on the PK and PD of IN-105 (Insulin Tregopil), an oral insulin; conducted in 3 sequential cohorts in an adaptive manner .

ELIGIBILITY:
Inclusion Criteria:

1. Patient should have an established diagnosis of T2DM per ADA 2013 criteria for at least 1 year prior to screening and are on metformin treatment for at least a month before screening.
2. Body mass index (BMI) of 18.5 to 40.00 kg/m2, both inclusive
3. Glycosylated hemoglobin (HbA1c) ≤ 9.5%.
4. Hemoglobin ≥9.0 g/dL.
5. No clinically significant abnormality in the ECG at screening.
6. Fasting plasma glucose levels less than 140 mg/dL at screening.
7. The patient should be ready to give a written and signed informed consent before starting any protocol-specific procedures.

Exclusion Criteria:

1. History of hypersensitivity to insulins or insulin analogues.
2. Evidence of the following (either due to improper diabetes control or due to secondary complications following diabetes).

   1. History of ≥2 episodes of severe hypoglycemia within 6 months before screening or history of hypoglycemia unawareness as judged by the investigator.
   2. History of ≥1 episodes of hyperglycemic hyperosmolar state or emergency room visits for uncontrolled diabetes leading to hospitalization in the 6 months prior to screening.
   3. History of limb amputation as a complication of diabetes during his/her lifetime or any vascular procedure during the 1 year prior to screening.
   4. History of diabetic foot or diabetic ulcers in the past 1 year prior to screening.
   5. History of severe form of neuropathy or cardiac autonomic neuropathy (determined when obtaining patient history).
3. Presence of any of the following:

   1. Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HBsAg) or hepatitis C infection at screening.
   2. Any clinically significant abnormality in the safety laboratory tests conducted at screening.
   3. Impaired hepatic function at screening [alanine transaminase (ALT) or aspartate aminotransferase (AST) value >2 times the upper limit of the reference range and/or serum bilirubin 1.5 times the upper limit of the reference range] which investigator considers clinically significant.
   4. Evidence of clinically significant chronic renal disease (e.g. nephrotic syndrome, diabetic nephropathy) as assessed by the investigator at screening
4. History or use of the following:

   1. Patients on OADs other than metformin for previous three months prior to screening.
   2. Patients who have received ≥14 consecutive days of oral, intravenous, or inhaled glucocorticoid therapy within the past 1 year or have received steroids by any route within 4 weeks immediately preceding screening visit (intra-nasal, intra ocular, and topical steroid use is allowed).
5. Receipt of another investigational drug in the 4 weeks prior to screening, or within 5 half-lives of the another investigational drug at screening visit (whichever is longer), or scheduled for another investigational drug during the current study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-last) will be assessed (Cohort 1) | from dosing time to 180 minutes post meal, extrapolated
  Area under the plasma concentration-time curve (AUC0-last; from dosing time to 180 minutes post meal, extrapolated) after single dose administration in the 30 ,20 and 10 minute pre-meal dosing groups
The maximum observed plasma drug concentration (Cmax) will be assessed (Cohort 1) | from dosing time to 180 minutes post meal
  The maximum observed plasma drug concentration after single dose administration (Cmax)
Glucose AUC0-t will be assessed (Cohort 1) | from dosing time to 180 minutes post meal
  Glucose AUC0-t [AUC both above and below the baseline values]
Glucose concentration (Cmin) will be assessed (Cohort 1) | from dosing time to 180 minutes post meal
  Minimum observed glucose concentration (Cmin)
Glucose concentration (Tmin) will be assessed (Cohort 1) | from dosing time to 180 minutes post meal
  Time of minimum observed glucose concentration (Tmin)
Area under the plasma concentration-time curve (AUC0-last) will be assessed (Cohort 2) | time of dosing to 180 minutes post dose,extrapolated
  Area under the plasma concentration-time curve (AUC0-last; time of dosing to 180 minutes post dose, extrapolated) after single dose administration in morning and afternoon in the 4, 5 and 6 h inter-meal interval groups.
The maximum observed plasma drug concentration (Cmax) will be assessed. (Cohort 2) | time of dosing to 180 minutes post dose
  The maximum observed plasma drug concentration after single dose administration (Cmax)
Glucose AUC0-t will be assessed (Cohort 2) | time of dosing to 180 minutes post dose
  Glucose AUC0-t [AUC both above and below the baseline values]
Glucose concentration (Cmin) will be assessed (Cohort 2) | time of dosing to 180 minutes post dose
  Minimum observed glucose concentration (Cmin)
Glucose concentration (Tmin) will be assessed (Cohort 2) | time of dosing to 180 minutes post dose
  Time of minimum observed glucose concentration (Tmin)
Area under the plasma concentration-time curve (AUC0-last) will be assessed (Cohort 3) | time of dosing to 180 minutes post dose,extrapolated
  Area under the plasma concentration-time curve (AUC0-last) for high-fat, high-fibre and ADA meal groups after single dose administration in morning and afternoon
The maximum observed plasma drug concentration (Cmax) will be assessed (Cohort 3) | time of dosing to 180 minutes post dose
  The maximum observed plasma drug concentration after single dose administration (Cmax)
Glucose AUC0-t will be assessed (Cohort 3) | time of dosing to 180 minutes post dose
  Glucose AUC0-t [AUC both above and below the baseline values]
Glucose concentration (Cmin) will be assessed. (Cohort 3) | time of dosing to 180 minutes post dose
  Minimum observed glucose concentration (Cmin)
Glucose concentration (Tmin) will be assessed. (Cohort 3) | time of dosing to 180 minutes post dose
  Time of minimum observed glucose concentration (Tmin)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Through study completion, approximately 3 months.
  An adverse event is any untoward medical event including hypoglycemia that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Rondon, M.D,JD, Principal Investigator — Elite Research Institute, 15705 NW 13th Avenue, Miami, Florida 33169

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khedkar A, Lebovitz H, Fleming A, Cherrington A, Jose V, Athalye SN, Vishweswaramurthy A. Pharmacokinetics and Pharmacodynamics of Insulin Tregopil in Relation to Premeal Dosing Time, Between Meal Interval, and Meal Composition in Patients With Type 2 Diabetes Mellitus. Clin Pharmacol Drug Dev. 2020 Jan;9(1):74-86. doi: 10.1002/cpdd.730. Epub 2019 Aug 7. PMID 31392840